CLINICAL TRIAL: NCT01683981
Title: Exercise Capacity and Quality of Life in Patients With Idiopathic Pulmonary Hypertension and Eisenmenger Syndrome Receiving Short Term Oral L-Citrulline Malate
Brief Title: Exercise Capacity and Quality of Life in Patients With PPH Receiving Short Term Oral L-Citrulline Malate
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masih Daneshvari Hospital (Other)
Responsible Party: Principal Investigator, babak sharif kashani, Head of Cardiology Department of NRITLD, Associate Professor, Masih Daneshvari Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: f-91-138
Record Dates: First submitted 2012-09-01; First posted 2012-09-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2012-09

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension; Eisenmenger Syndrome
Keywords: Idiopathic Pulmonary Arterial Hypertension; Eisenmenger Syndrome; Exercise Capacity; Quality of Life
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Eisenmenger Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-Citrulline, Exercise Capacity (Experimental): L-Citrulline malate, 1gr, oral, divided 3 times a day,for 2 weeks
  Interventions: Drug: L-Citrulline Malate

INTERVENTIONS:
Drug: L-Citrulline Malate — 3 gr per day, oral, for 2 weeks
  Other Names: Stimol

SUMMARY:
Due to vasodilatory properties of the NO, one of the therapeutic approaches for IPAH is oral use of nitric oxide precursors (10). Efficacy of L-arginine is well-documented in the current literature but there is paucity of data with regard to L-citrulline- malate. Hence, this study will evaluate therapeutic efficacy of L-citrulline- malate in two categories of patients with pulmonary hypertension (IPAH, and Eisenmeger syndrome). This randomized clinical trial utilizes 6-minute walk, pro BNP levels and the echocardiographic indexes an indicator of functional improvement of the patients.

DETAILED DESCRIPTION:
Pulmonary vascular tone is maintained by the action of vasoprotective compounds including nitric oxide (NO)(1).NO can be synthesized endogenously in the body via L-arginine and NOS-independent mechanism from the anion nitrite (NO2-)(2,3).Nitric oxide (NO) causes cyclic guanosine monophosphate-mediated vasodilatation of the pulmonary vasculature. Endogenous NO is also produced from the metabolism of citrulline; an amino acid generated by the urea cycle (4). NO is critical for normal development of the pulmonary vasculature and loss of this vasodilator factor and subsequent endothelial dysfunction is proposed as one of the possible explanations for development of pulmonary hypertension (1).

From a clinical standpoint, pulmonary hypertension is a common complication of chronic obstructive pulmonary disease (COPD).Its presence is associated with shorter survival and worse clinical outcome. In a setting of COPD, pulmonary hypertension tends to be of moderate severity and progresses slowly. Recent investigations have demonstrated endothelial dysfunction and changes in the expression of endothelial-derived mediators that regulate vascular tone and cell growth in the pulmonary arteries of patients with mild disease(5). Pulmonary vascular involvement from congenital heart disease like Eisenmeger syndrome is another important category of patients with PAH. In this congenital disease pulmonary vascular involvement follows a period in which pulmonary resistance is low and pulmonary blood flow is high (6, 7, 8). Finally, Idiopathic pulmonary hypertension (IPAH) is the third category of these patients. IPAH has unknown etiology and is characterized by progressive obliteration of small and medium size pulmonary arteries; elevation in pulmonary arterial pressure, and an increase in pulmonary vascular resistance. Presence of these pathologies eventually leads to right heart failure and death (9).

ELIGIBILITY:
Inclusion Criteria:

* all patients less than 70 years old,
* patients with a six-minute walking distance of more than 100 meters (m),
* a mean pulmonary arterial pressure (PAP) ≥ 25 mmHg at rest as assessed by right heart catheterization(RHC) (11,12).

Exclusion Criteria:

* all patients more than 70 years old,
* patients with a six-minute walking distance of less than 100 meters (m), active pulmonary or extra pulmonary infection,
* serious coronaropathy and/ or ventricular dysfunction,
* significant renal illness and/or hepatitis,
* detected immunosuppressive illnesses,
* carrier of known neoplasias,
* pregnancy,
* lack of family support,
* psychosocial problems,
* drug or alcohol abuse, and
* noncompliance with established medical protocol.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
the change in exercise capacity | 2 weeks
  The primary measure of efficacy was the change in exercise capacity, as measured by the total distance walked in six minutes, from baseline to week 2. (15)

SECONDARY OUTCOMES:
changes in mean pulmonary-artery pressure | 2 weeks
  changes in mean pulmonary-artery pressure from baseline to week 2.

OTHER OUTCOMES:
change in the quality of life | 2 weeks
  change in the quality of life from baseline to week 2

CONTACTS AND LOCATIONS:
Overall Officials: babak sharif kashani, cardiologist, Principal Investigator — Lung Transplantation Research Center, National Research Institute of Tuberculosis and Lung Disease (NRITLD), Shahid Beheshti University of Medical Science, Tehran, Iran.; Paritash Tahmaseb pour, MD, Principal Investigator — MD
Locations (1):
- MasihDH, Tehran, Iran